CLINICAL TRIAL: NCT06974188
Title: AI-Powered CURAᵀᴹ Application for Identifying At-Risk Pregnancies in Obstetric Management: A Randomized Controlled Trial (CURAte)
Brief Title: AI-Powered CURAᵀᴹ Application for Identifying At-Risk Pregnancies in Obstetric Management
Acronym: CURAte
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Collaborators: National University of Singapore (Other); National University of Singapore, Saw Swee Hock School of Public Health (Unknown); Agency for Science, Technology and Research (A*STAR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Screening
Other Study IDs: 2024-3832
Record Dates: First submitted 2025-04-29; First posted 2025-05-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2024-11

CONDITIONS: High-risk Pregnancy; Pregnancy; Antenatal Health
Keywords: Machine-learning; Artificial Intelligence; Antenatal Risk Stratification; Software as a Medical Device; Machine Learning Algorithm; Pregnancy Complications; Neonatal Complications; Pregnancy outcomes; Obstetric complications; Antenatal care
MeSH Terms: conditions — Pregnancy Complications

STUDY DESIGN:
Intervention Model Description: The study employs a two parallel arm, single-blinded, pragmatic randomised controlled trial design. In this design, pregnant women will be randomly assigned in a 1:1 ratio to an AI-assisted risk categorization approach or the current manual risk stratification method.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AI-risk stratification arm (Experimental): During their first trimester antenatal visit, participants will be risk stratified by clinicians with the assistance of AI. The risk prediction of 'high risk' or 'low risk' will be immediately made known to the clinician during the visit.
  Similarly, during the 31 -34 weeks visit following release of oral glucose tolerance test and growth scan results, participants will be risk stratified by clinicians again with the assistance of AI.
  Interventions: Other: AI-risk Stratification
- Non-AI arm (Current Risk Stratification) (No Intervention): During their first trimester antenatal visit, participants will be risk stratified by both clinicians alone and with the assistance of AI. However, the risk prediction of 'high risk' or 'low risk' will not be disclosed to the clinician at all. It will only be revealed to the study investigators at the end of the study.
  Similarly, during the 31 -34 weeks visit following release of oral glucose tolerance test and growth scan results, participants will be risk stratified by clinicians again with and without the assistance of AI. However, the risk prediction of 'high risk' or 'low risk' will not be disclosed to the clinician at all. It will only be revealed to the study investigators at the end of the study.
  Clinicians will use their own judgement as to the risk of the participants' pregnancies. They have to adhere to the same specific 'high-risk' and 'low-risk' management protocol.

INTERVENTIONS:
Other: AI-risk Stratification — With the results being disclosed as 'high-risk' or 'low-risk' in the experimental arm, clinicians have to adhere to a specific 'high-risk' and 'low-risk' management protocol for participants.
  Arms: AI-risk stratification arm

SUMMARY:
It is important to identify high pregnancies early through screening so that appropriate care and intervention may be instituted. An AI-assisted risk categorisation approach may be advantageous compared with traditional means of screening. The purpose of this study is to determine if the adoption of an AI-assisted approach in general pregnancy risk screening will improve the accuracy of antenatal risk categorization into high- and low- risk pregnancy groups, ultimately resulting in fewer poor maternal and fetal/neonatal outcomes.

DETAILED DESCRIPTION:
High-risk pregnancies refer to pregnancies at risk of an adverse maternal outcomes (e.g., gestational diabetes, pre-eclampsia) or fetal/neonatal (e.g. preterm birth, still birth, hypoxic-ischemic encephalopathy). In most healthcare facilities, antenatal care is delivered through a general obstetric clinic. The initial screening of risk is guided by the patient's past medical history, past obstetric history for multigravida patients, and the individual provider's knowledge, which may vary across years of experience in the field. Therefore, the triaging of patients into appropriate antenatal care pathways is inconsistent and often inaccurate. AI technology, particularly Machine Learning (ML) has potential to develop predictive models that are able to segregate low-risk from high-risk pregnancies using complex interactions and relationships. The investigators propose a novel AI-assisted risk stratification model in pregnancy that can help to overcome the current gaps. The AI model considers maternal history and simple biophysical measurements performed in pregnancy.

The primary objective of the CURAte trial is to compare the composite incidence of maternal and fetal/neonatal adverse outcomes between participants who were randomised to the AI-assisted risk stratification intervention arm and participants who were randomised to the no-AI assisted control arm. The secondary objective is to test the feasibility and acceptability of an AI-assisted antenatal risk stratification approach in a real-life patient-care system.

The study will adopt a parallel arm single-blinded, pragmatic randomised controlled trial design. Women presenting at the subsidised antenatal clinics in the first trimester will be approached and assessed for eligibility. A total of 1444 participants (722 in each arm) will be recruited in this study. All participants will be randomised via block randomisation in a 1:1 ratio into two groups (AI-assisted arm versus non-AI assisted arm (standard of care)) which will be done through an electronic programme prepared by the trial statistician. Enrolled participants will be required to complete a questionnaire about their sociodemographic, obstetric and medical history on the FormSG platform prior to consultation with the clinician. The AI-assisted risk stratification will be deployed twice in each participant's pregnancy- at the first trimester visit before 13 weeks' and 6 days' gestation, followed by after the results of the oral glucose tolerance test and third trimester growth scan are available, usually between 31- and 33-weeks' gestation. The results of the AI-assisted risk stratification will not be disclosed in the no-AI intervention arm, until the end of the study. Other study data (i.e. pre-specified study outcomes) will be extracted from medical records at or after 6 weeks from delivery (or at the end of pregnancy) to assess the primary and secondary outcomes.

The primary analysis will be conducted on an intention-to-treat basis, for the binary primary composite outcome of maternal/fetal and neonatal morbidity and mortality. For improved precision, a further multiple regression adjusting for factors known to be prognostic of pregnancy and neonatal outcomes including maternal age, BMI, parity, ethnicity will also be conducted. The investigators' proposed new AI-assisted screening model will address the current gaps in the stratification approach and improve the clinical relevance of antenatal screening in the long run, with downstream positive impact on maternal and neonatal well-being, as well as potential cost savings to the healthcare system. By testing this AI-assisted model in an actual clinical setting in a public healthcare institution, the investigators will be able to identify challenges relating to real-world logistics and enablers for translating this digital innovation into clinical practice. The investigators can use the findings to elicit specific modifications to both the AI-assisted model workflow and CuraTM application, ultimately optimising the future implementation as well as acceptability and uptake amongst healthcare providers and pregnant women.

ELIGIBILITY:
Inclusion Criteria:

* Age: 21 years old to 50 years old
* Singleton Pregnancy
* No more than 13 weeks' and 6 days' gestation at recruitment
* Able to provide written, informed consent

Exclusion Criteria:

* Not proficient in the English language (AI intervention is only available in English at this stage)

Ages: 21 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1700 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
The number and proportion of cases displaying any one of the following outcomes listed below (composite): | At Delivery (Birth)
  Presented as a relative risk (RR) with 95% CI, with and without stratification for parity, ethnicity and BMI.
  (i) Maternal
  * Postpartum haemorrhage more than/equal to 1000ml or requiring blood product transfusion
  * Eclampsia/severe eclampsia (blood pressure SBP>160mmHg or diastolic >110mmHg and/or significant end-organ damage which can include signs of liver or kidney impairment, low platelet count, fluid in the lungs or new-onset headache/visual disturbances)
  * ICU or HDU admission (excluding those who are admitted for precautionary monitoring)
  * Unplanned hysterectomy
  * Uterine rupture (symptomatic full thickness rupture)
  * Venous thromboembolism proven radiologically
  * Maternal mortality
  (ii) Neonatal:
  * Apgar scores <7 at 5 minutes or less than/equal to 4 at 10 minutes
  * Respiratory distress requiring mechanical ventilation or surfactant treatment
  * Hypoxic ischaemic encephalopathy (HIE, any grade)
  * neonatal death (within 28 days of birth)/
  * intrauterine demise
In addition, these outcomes will be reported individually: | At Delivery (Birth)
  Number and proportion, RR and 95% CI for each of the following:
  * Postpartum haemorrhage more than/equal to 1000ml or requiring blood product transfusion as well as mean difference in blood loss
  * Eclampsia/severe eclampsia (blood pressure SBP>160mmHg or diastolic >110mmHg and/or significant end-organ damage which can include signs of liver or kidney impairment, low platelet count, fluid in the lungs or new-onset headache/visual disturbances) as well as difference in gestational age of onset or diagnosis with and without adjustment for important covariates
  * ICU or HDU admission (excluding those who are admitted for precautionary monitoring)
  * Maternal mortality as well as cause of death
  * Respiratory distress requiring mechanical ventilation or surfactant treatment as well as aetiology for RDS
  * Hypoxic ischaemic encephalopathy (HIE, any grade)
  * Neonatal death (within 28 days of birth)
  * Intrauterine demise

SECONDARY OUTCOMES:
To test the feasibility of an AI-assisted antenatal risk stratification approach in a real-life patient-care system - Quantitative; Mean Differences | At baseline visit (first trimester antenatal visit)
  * Mean differences or categorically-determined outcomes of time taken for each participant to complete the questionnaire
  * Mean differences or categorically-determined outcomes of time taken for each consultation with the clinician to complete the questionnaire and launch AI
To test the feasibility of an AI-assisted antenatal risk stratification approach in a real-life patient-care system - Qualitative | At baseline visit (first trimester antenatal visit)
  * Qualitative Feedback to determine acceptability by participants and clinicians
  * Clinicians' actions in response to the AI results for all cases: low, high, undisclosed to assess mechanisms in which AI influences clinicians' decision- making
To test the feasibility of an AI-assisted antenatal risk stratification approach in a real-life patient-care system - Quantitative; Number | At baseline visit (first trimester antenatal visit)
  • Number of (potential) participants screened and recruited per antenatal clinic session

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Li, MRCOG, MPH, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Rivera SC, Liu X, Chan AW, Denniston AK, Calvert MJ; SPIRIT-AI and CONSORT-AI Working Group. Guidelines for clinical trial protocols for interventions involving artificial intelligence: the SPIRIT-AI Extension. BMJ. 2020 Sep 9;370:m3210. doi: 10.1136/bmj.m3210. PMID 32907797
- [Background] Malacova E, Tippaya S, Bailey HD, Chai K, Farrant BM, Gebremedhin AT, Leonard H, Marinovich ML, Nassar N, Phatak A, Raynes-Greenow C, Regan AK, Shand AW, Shepherd CCJ, Srinivasjois R, Tessema GA, Pereira G. Stillbirth risk prediction using machine learning for a large cohort of births from Western Australia, 1980-2015. Sci Rep. 2020 Mar 24;10(1):5354. doi: 10.1038/s41598-020-62210-9. PMID 32210300
- [Background] Jhee JH, Lee S, Park Y, Lee SE, Kim YA, Kang SW, Kwon JY, Park JT. Prediction model development of late-onset preeclampsia using machine learning-based methods. PLoS One. 2019 Aug 23;14(8):e0221202. doi: 10.1371/journal.pone.0221202. eCollection 2019. PMID 31442238
- [Background] Arabi Belaghi R, Beyene J, McDonald SD. Prediction of preterm birth in nulliparous women using logistic regression and machine learning. PLoS One. 2021 Jun 30;16(6):e0252025. doi: 10.1371/journal.pone.0252025. eCollection 2021. PMID 34191801
- [Background] Bhutta ZA, Das JK, Bahl R, Lawn JE, Salam RA, Paul VK, Sankar MJ, Blencowe H, Rizvi A, Chou VB, Walker N; Lancet Newborn Interventions Review Group; Lancet Every Newborn Study Group. Can available interventions end preventable deaths in mothers, newborn babies, and stillbirths, and at what cost? Lancet. 2014 Jul 26;384(9940):347-70. doi: 10.1016/S0140-6736(14)60792-3. Epub 2014 May 19. PMID 24853604
- [Background] Gosavi A, Amin Z, Carter SWD, Choolani MA, Fee EL, Milad MA, Jobe AH, Kemp MW. Antenatal corticosteroids in Singapore: a clinical and scientific assessment. Singapore Med J. 2024 Sep 1;65(9):479-487. doi: 10.4103/SINGAPOREMEDJ.SMJ-2022-014. Epub 2022 Oct 6. PMID 36254928
- [Background] Hewage S, Audimulam J, Sullivan E, Chi C, Yew TW, Yoong J. Barriers to Gestational Diabetes Management and Preferred Interventions for Women With Gestational Diabetes in Singapore: Mixed Methods Study. JMIR Form Res. 2020 Jun 30;4(6):e14486. doi: 10.2196/14486. PMID 32602845
- [Background] Phibbs CM, Kozhimannil KB, Leonard SA, Lorch SA, Main EK, Schmitt SK, Phibbs CS. A Comprehensive Analysis of the Costs of Severe Maternal Morbidity. Womens Health Issues. 2022 Jul-Aug;32(4):362-368. doi: 10.1016/j.whi.2021.12.006. Epub 2022 Jan 12. PMID 35031196
- [Background] Chi C, Pang D, Aris IM, Teo WT, Li SW, Biswas A, Yong EL, Chong YS, Tan K, Kramer MS. Trends and predictors of cesarean birth in Singapore, 2005-2014: A population-based cohort study. Birth. 2018 Dec;45(4):399-408. doi: 10.1111/birt.12341. Epub 2018 Feb 17. PMID 29453821
- [Background] Fink DA, Kilday D, Cao Z, Larson K, Smith A, Lipkin C, Perigard R, Marshall R, Deirmenjian T, Finke A, Tatum D, Rosenthal N. Trends in Maternal Mortality and Severe Maternal Morbidity During Delivery-Related Hospitalizations in the United States, 2008 to 2021. JAMA Netw Open. 2023 Jun 1;6(6):e2317641. doi: 10.1001/jamanetworkopen.2023.17641. PMID 37347486